CLINICAL TRIAL: NCT04430634
Title: An Open-Label, Randomized, Crossover Study to Assess Nicotine Uptake, Tobacco-Related Biomarkers of Exposure, Biomarkers of Potential Harm, and Puff Topography With Use of mybluTM Electronic Cigarettes in Adult Smokers
Brief Title: A Study to Evaluate Nicotine Uptake and Biomarkers in Smokers Using mybluTM Electronic Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fontem US LLC (Industry)
Collaborators: Fontem Ventures BV (Industry)
Responsible Party: Sponsor
Organization: Fontem Ventures BV (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: CA22749
Record Dates: First submitted 2020-06-10; First posted 2020-06-12 (Actual); Results first posted 2021-06-07 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-05

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- ABDC (Experimental): Subjects use MybluTM e-cigarette product variant A (2.4 % nicotine) ad libitum for 2 days, then switch to use variant B (3.6% nicotine) for 2 days, then D (4.0% nicotine) for 2 days and then C (2.5% nicotine) for 2 days. A washout period of 12 hours product abstinence is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
  Interventions: Other: Myblu variant A; Other: Myblu variant B; Other: Myblu variant C; Other: Myblu variant D
- BCAD (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu variant A; Other: Myblu variant B; Other: Myblu variant C; Other: Myblu variant D
- CDBA (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu variant A; Other: Myblu variant B; Other: Myblu variant C; Other: Myblu variant D
- DACB (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu variant A; Other: Myblu variant B; Other: Myblu variant C; Other: Myblu variant D
- EFHG (Experimental): Subjects use MybluTM e-cigarette product variant E (3.6 % nicotine) ad libitum for 2 days, then switch to use variant F (2.4% nicotine) for 2 days, then H (3.6% nicotine) for 2 days and then G (4.0% nicotine) for 2 days. A washout period of 12 hours product abstinence is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
  Interventions: Other: Myblu variant E; Other: Myblu variant F; Other: Myblu variant G; Other: Myblu variant H
- FGEH (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu variant E; Other: Myblu variant F; Other: Myblu variant G; Other: Myblu variant H
- GHFE (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu variant E; Other: Myblu variant F; Other: Myblu variant G; Other: Myblu variant H
- HEGF (Experimental): Same as previous arm, but in a different randomization order.
  Interventions: Other: Myblu variant E; Other: Myblu variant F; Other: Myblu variant G; Other: Myblu variant H

INTERVENTIONS:
Other: Myblu variant A — Use of Myblu e-cigarette with flavor A 2.4% nicotine
  Arms: ABDC; BCAD; CDBA; DACB
Other: Myblu variant B — Use of Myblu e-cigarette with flavor B 3.6% nicotine
  Arms: ABDC; BCAD; CDBA; DACB
Other: Myblu variant C — Use of Myblu e-cigarette with flavor C 2.5% nicotine
  Arms: ABDC; BCAD; CDBA; DACB
Other: Myblu variant D — Use of Myblu e-cigarette with flavor D 4.0% nicotine
  Arms: ABDC; BCAD; CDBA; DACB
Other: Myblu variant E — Use of Myblu e-cigarette with flavor E 3.6% nicotine
  Arms: EFHG; FGEH; GHFE; HEGF
Other: Myblu variant F — Use of Myblu e-cigarette with flavor F 2.4% nicotine
  Arms: EFHG; FGEH; GHFE; HEGF
Other: Myblu variant G — Use of Myblu e-cigarette with flavor G 4.0% nicotine
  Arms: EFHG; FGEH; GHFE; HEGF
Other: Myblu variant H — Use of Myblu e-cigarette with flavor H 3.6% nicotine
  Arms: EFHG; FGEH; GHFE; HEGF

SUMMARY:
This study evaluates the overall performance of the currently-marketed MybluTM e-cigarette device and pods, as assessed by nicotine uptake, exposure to smoke constituents, safety and consumer satisfaction, over 8 days. The study is designed as an open-label, randomized study in adult smokers.

Subjects are invited to participate to a second part of the study, for 5 additional days, to compare the use of MybluTM to the use of subject's usual brand combustible cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* smoking an average of at least 10 manufactured combustible cigarettes per day for at least 12 months prior to Screening
* tested positive for urine cotinine (≥ 200 ng/mL) at Screening
* exhaled carbon monoxide > 10 ppm (parts per million) at Screening

Exclusion Criteria:

* relevant illness history
* relevant medication use
* body mass index (BMI) > 40 kg/m2 or < 18 kg/m2 at Screening
* allergy to propylene glycol or glycerin
* use of nicotine-containing products other than manufactured combustible cigarettes within 14 days prior to Check-in
* use of any prescription smoking cessation treatments within 3 months prior to Check-in
* smokers who draw smoke from the cigarette into the mouth and throat but do not inhale
* planning to quit smoking during the study
* female subjects who are pregnant, lactating, or intend to become pregnant

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Morris P, McDermott S, Chapman F, Verron T, Cahours X, Stevenson M, Thompson J, Chaudhary N, O'Connell G. Reductions in biomarkers of exposure to selected harmful and potentially harmful constituents following exclusive and partial switching from combustible cigarettes to myblu electronic nicotine delivery systems (ENDS). Intern Emerg Med. 2022 Mar;17(2):397-410. doi: 10.1007/s11739-021-02813-w. Epub 2021 Aug 26. PMID 34435305

RESULTS

PARTICIPANT FLOW:
Groups:
- ABDC: Subjects use MybluTM e-cigarette product variant A (2.4 % nicotine) ad libitum for 2 days, then switch to use variant B (3.6% nicotine) for 2 days, then D (4.0% nicotine) for 2 days and then C (2.5% nicotine) for 2 days. A 12-hour washout period is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
- BCAD; CDBA; DACB; FGEH; GHFE; HEGF: Same as previous but in a different randomization order
- EFHG: Subjects use MybluTM e-cigarette product variant E (3.6 % nicotine) ad libitum for 2 days, then switch to use variant F (2.4% nicotine) for 2 days, then H (3.6% nicotine) for 2 days and then G (4.0% nicotine) for 2 days. A 12-hour washout period is observed between product variants. For each product variant, in the morning of the second product use day, a controlled product use session is performed (10 puffs taken at 30-second intervals, with puffs 3 seconds in duration).
Period: Overall Study
Arm/Group | ABDC | BCAD | CDBA | DACB | EFHG | FGEH | GHFE | HEGF
Started | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5
Completed | 5 | 5 | 5 | 4 | 5 | 5 | 4 | 5
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABDC | BCAD | CDBA | DACB | EFHG | FGEH | GHFE | HEGF | Total
Number analyzed (Participants) | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 5 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (15.28) | 38.6 (14.03) | 47.6 (8.73) | 37.8 (10.76) | 44.6 (10.88) | 41.6 (11.19) | 43.0 (11.51) | 47.2 (12.58) | 43.3 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 2 | 1 | 2 | 1 | 1 | 4 | 16
  Male | 2 | 3 | 3 | 4 | 3 | 4 | 4 | 1 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 5 | 5 | 5 | 4 | 5 | 5 | 5 | 5 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body mass index
  kg/m^2 | 25.8 (4.5) | 29.3 (2.1) | 29.4 (5.5) | 29.2 (4.3) | 26.4 (7.3) | 25.3 (3.3) | 28.2 (3.7) | 27.5 (3.3) | 27.6 (4.4)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Nicotine Concentration in Blood
Description: Maximum nicotine concentration in blood (Cmax)
Time Frame: 180 minutes following the start of the controlled product use session on Day 2 (12 measurements over the period)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- Product Variant A: MyBlu e-cigarette variant A (2.4% nicotine)
- Product Variant B: MyBlu e-cigarette variant B (3.6% nicotine)
- Product Variant C: MyBlu e-cigarette variant C (2.5% nicotine)
- Product Variant D: MyBlu e-cigarette variant D (4.0% nicotine)
- Product Variant E: MyBlu e-cigarette variant E (3.6% nicotine)
- Product Variant F: MyBlu e-cigarette variant F (2.4% nicotine)
- Product Variant G: MyBlu e-cigarette variant G (4.0% nicotine)
- Product Variant H: MyBlu e-cigarette variant H (3.6% nicotine)
Arm/Group | Product Variant A | Product Variant B | Product Variant C | Product Variant D | Product Variant E | Product Variant F | Product Variant G | Product Variant H
Number analyzed (Participants) | 19 | 18 | 19 | 18 | 18 | 19 | 19 | 18
ng/mL | 3.6 (91.6) | 5.3 (109.6) | 4.0 (113.5) | 5.3 (106.4) | 6.5 (135.7) | 4.6 (143.4) | 8.0 (99.6) | 9.3 (95.8)

2. Primary Outcome: Concentration of Carboxyhemoglobin in Blood
Description: Change from baseline in the concentration of carboxyhemoglobin (COHb) in whole blood.
Time Frame: Baseline and 8 days
Population: The arms are combined into one group, because the aim was to compare biomarkers in all participants who use any e-cigarette variant, to the value at baseline (when they were smoking conventional cigarettes). Data is missing for 2 participants at the 8 days timepoint.
Measure: Mean (Standard Deviation); unit: % saturation
Groups:
- Exclusive MyBlu E-cigarette Use: Subjects who used any MyBlu e-cigarette variant for 8 days (all subjects who completed Part 1 of the study)
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 39
% saturation
  Baseline value | 7.7 (2.1)
  Change from baseline: number analyzed (Participants) | 37
  Change from baseline | -6.25 (2.06)

3. Primary Outcome: Amount of 4-(Methylnitrosamino)-1-(3-pyridyl)-1-butanol in Urine in 24 Hours
Description: Change from baseline in the amount of 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanol (NNAL), a biomarker of exposure to 4-(methylnitrosamino)-1-(3-pyridyl)-1-butanone (NNK), excreted in urine during 24 hours (creatinine adjusted).
Time Frame: Baseline and 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/g creatinine
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 39
ng/g creatinine
  Baseline value | 345.4 (252.3)
  Change from baseline: number analyzed (Participants) | 37
  Change from baseline | -262.8 (205.1)

4. Primary Outcome: Amount of 3-hydroxypropylmercapturic Acid in Urine in 24 Hours
Description: Change from baseline in the amount of 3-hydroxypropylmercapturic acid (3-HPMA), a biomarker of exposure to acrolein, excreted in urine during 24 hours (creatinine adjusted).
Time Frame: Baseline and 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/g creatinine
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 39
ug/g creatinine
  Baseline value | 1242.2 (536.0)
  Change from baseline: number analyzed (Participants) | 37
  Change from baseline | -1097.1 (522.2)

5. Primary Outcome: Amount of S-phenyl Mercapturic Acid in Urine in 24 Hours
Description: Change from baseline in the amount of S-phenyl mercapturic acid (S-PMA), a biomarker of exposure to benzene, excreted in urine during 24 hours (creatinine adjusted).
Time Frame: Baseline and 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ug/g creatinine
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 39
ug/g creatinine
  Baseline value | 5.9 (4.2)
  Change from baseline: number analyzed (Participants) | 37
  Change from baseline | -5.9 (4.1)

6. Secondary Outcome: Level of White Blood Cells
Description: The change from baseline in the level of white blood cells, a biomarker of potential harm.
Time Frame: Baseline and 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 39
cells*10^9/L
  Baseline value | 7.5 (1.7)
  Change from baseline: number analyzed (Participants) | 37
  Change from baseline | -0.4 (1.1)

7. Secondary Outcome: Spirometry: Forced Expiratory Volume in 1 Second
Description: Forced expiratory volume in 1 second (FEV1) measurement conducted in accordance with the 2005 American Thoracic Society / European Respiratory Society Joint Task Force on the standardization of spirometry, with subject in a sitting position following at least 15 minutes of rest and at least 1 hour from the last product use.
Time Frame: Baseline and 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
L
  Baseline value | 2.9 (1.2)
  8 days timepoint: number analyzed (Participants) | 36
  8 days timepoint | 3.2 (0.9)

8. Secondary Outcome: Spirometry: Forced Vital Capacity
Description: Forced vital capacity (FVC) measurement conducted in accordance with the 2005 American Thoracic Society / European Respiratory Society Joint Task Force on the standardization of spirometry, with subject in a sitting position following at least 15 minutes of rest and at least 1 hour from the last product use.
Time Frame: Baseline and 8 days
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Exclusive MyBlu E-cigarette Use
Number analyzed (Participants) | 38
L
  Baseline value | 3.8 (1.5)
  8 days timepoint: number analyzed (Participants) | 36
  8 days timepoint | 4.2 (1.2)

9. Secondary Outcome: Subjective Measure: Urge to Smoke
Description: Urge to smoke score: Subjects answer the following question "How strong is your urge to smoke right now?" using a visual analogue scale (VAS). The scale ranges from "Not at all", given a score of 0, to "Extremely", given a score of 100, after ad libitum use of the product.
Time Frame: 8 days
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Product Variant A | Product Variant B | Product Variant C | Product Variant D | Product Variant E | Product Variant F | Product Variant G | Product Variant H
Number analyzed (Participants) | 19 | 19 | 19 | 19 | 19 | 19 | 20 | 19
score on a scale | 70.4 (18.7) | 67.8 (24.8) | 67.2 (21.7) | 63.7 (22.1) | 62.0 (31.6) | 56.2 (34.4) | 62.9 (32.1) | 63.0 (29.4)

ADVERSE EVENTS:
Time Frame: 9 days
Arm/Group | Product Variant A | Product Variant B | Product Variant C | Product Variant D | Product Variant E | Product Variant F | Product Variant G | Product Variant H
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/20 | 0/19 | 0/19 | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/19 | 0/19 | 0/20 | 0/19 | 0/19 | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/19 | 4/19 | 3/19 | 2/20 | 3/19 | 2/19 | 0/20 | 3/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Product Variant A (N=19) | Product Variant B (N=19) | Product Variant C (N=19) | Product Variant D (N=20) | Product Variant E (N=19) | Product Variant F (N=19) | Product Variant G (N=20) | Product Variant H (N=20)
Dizziness (Nervous system disorders) | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eyelid pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Swelling of eyelid (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT04430634/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-20): https://cdn.clinicaltrials.gov/large-docs/34/NCT04430634/SAP_001.pdf